CLINICAL TRIAL: NCT07057999
Title: Effects of the MIND Diet on Fatigue, Quality of Life, and Brain Fog in Patients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Investigation of the Effect of the MIND Diet on Disease Symptoms in Patients With MS
Acronym: MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betul Uner (Other)
Responsible Party: Sponsor-Investigator, Betul Uner, Lecturer, MSc, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Decision number 2025/643
Record Dates: First submitted 2025-06-18; First posted 2025-07-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis; Diet Therapy; Body Composition; Randomised Controlled Trial; Brain Fog; Fatigue Syndrome, Chronic; Quality of Life (QOL)
MeSH Terms: conditions — Multiple Sclerosis; Mental Fatigue; Fatigue Syndrome, Chronic | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The planned study will be conducted in the Neurology Outpatient Clinic of Muğla Education and Research Hospital and will use a parallel-group, open-label, randomized controlled trial design. Randomization, where each participant has an equal chance of being assigned to the intervention group, is an effective way to prevent the risk of selection bias. Block randomization will be used to determine the intervention and control groups in the planned study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): MIND Diet Program
  Interventions: Behavioral: MIND Diet (Mediterranean-DASH Intervention for Neurodegenerative Delay)
- control group (Active Comparator): Traditional Healthy Nutrition Program
  Interventions: Behavioral: Traditional healthy nutrition program specific to Turkey

INTERVENTIONS:
Behavioral: MIND Diet (Mediterranean-DASH Intervention for Neurodegenerative Delay) — The MIND diet consists of 15 components. While the first 10 of the components are considered healthy for the brain, the last 5 are considered unhealthy. The MIND diet portion and consumption frequency recommendations are as follows; olive oil consumption ≥ 48 g/day; oil seeds and nuts ≥ 5 servings/week; green leafy vegetables ≥1 serving/day; cooked vegetables ≥1 serving/day; whole grains ≥3 servings/day; legumes 3 servings/week; red fruits such as blueberries and strawberries ≥2 servings/week; poultry ≥2 servings/week; fish and seafood ≥1 serving week; red wine 1 glass/day; red meat ≤4 servings/week; butter ≤10 g/day; bakery products <5 servings/week; fast food <1 serving/week. Patients assigned to this group will be given a diet program based on isocaloric, MIND diet principles, which they will be asked to follow for 12 weeks.
  Other Names: MIND diet; DASH; Mediterranean diet
  Arms: intervention group
Behavioral: Traditional healthy nutrition program specific to Turkey — There are no prohibited foods in the traditional Türkiye-specific nutrition recommendations included in the TÜBER 2022 report, but there are foods that are recommended to be restricted or increased. According to the healthy nutrition program, 3 portions/day from the milk and dairy products (milk, yogurt, kefir, cheese) group; 2.5-3 portions/day from the meat, chicken, fish, eggs, legumes, oilseeds and nuts group; 2.5-4 portions/day from the vegetable group; 2-3 portions/day from the fruit group; 3-7 portions/day from the bread and cereal group; 3-4 portions/day from the fat group and finally, simple sugar consumption is recommended as a maximum of 10% of total energy. An isocaloric diet will be prepared according to the body composition and eating habits of the patients and they will be asked to follow it for 12 weeks.
  Arms: control group

SUMMARY:
The planned parallel group, randomized controlled study design will be used to determine the effects of the MIND diet applied to MS patients on fatigue, quality of life, technological function and brain fog and to contribute to the scientific literature. This study document will also determine the scope of the MIND diet for MS details. The regular questions it aims to answer are as follows:

* Is the MIND diet applied to MS treatments effective on quality of life compared to traditional healthy nutrition?
* Is the MIND diet applied to MS treatments effective on fatigue compared to traditional healthy nutrition therapy?
* Is the MIND diet applied to MS treatments effective on brain fog compared to traditional healthy nutrition therapy?

In this study, the MIND diet will be controlled with a traditional healthy nutrition program specific to Türkiye to evaluate the effect of the MIND diet on MS disease.

Participants:

* Adhere to your specially prepared diet for 3 months
* Participate in online meetings with researchers every week to check compliance with the diets
* Visit the hospital for a check-up at the end of 3 months The collected study data will be analyzed in a computer environment using the Statistical Package for Social Sciences (IBM, SPSS, version 29.0) software, and p<0.05 is accepted as the significance level.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is defined as an autoimmune disease of the central nervous system that causes myelin loss and axonal damage and is characterized by inflammation. MS can also occur as acute optic neuritis, brainstem syndrome, pyramidal system demyelination and/or spinal cord syndromes. In addition to neurological symptoms such as vision loss, weakness, numbness, difficulty walking and dysesthesia due to demyelination occurring during the formation of the disease, atypical symptoms such as fatigue, depression and cognitive disorders are also observed. Although early and accurate diagnosis of MS is essential, diagnosis is based on the presence of clinical symptoms and findings on magnetic resonance imaging (MRI), which is highly sensitive in detecting characteristic central nervous system lesions. McDonald 2017 criteria are used in the diagnosis of the disease.

There are four clinically defined types of the disease. The types of MS are; relapsing-remitting MS, which constitutes approximately 85% of cases, primary progressive MS, which constitutes 10-20% of cases, secondary progressive MS, and clinically isolated syndrome. In patients with relapsing-remitting MS, the transmission of nerve impulses is affected during relapses, while the course of the disease and symptoms tend to improve or improve during remission. When relapses increase, progressive neural dysfunction occurs, and when remission is not achieved, progressive neurological damage occurs. This condition is defined as secondary progressive MS. In order to diagnose primary progressive MS, the disability status that continues for at least one year must be progressive. However, distinguishing between primary progressive MS and secondary progressive MS is often challenging. Although the course of the disease varies greatly depending on the type, many people develop irreversible disability, and MS continues to be the leading cause of neurological disability in young adults. The disability levels of individuals with MS are determined by the Expanded Disability Status Scale (EDSS). EDSS is a scale used worldwide in the evaluation and follow-up of neurological examinations of patients. The EDSS score ranges from 0 to 10. A score of 0 means "normal neurological examination, no disability", while a score of 10 means "death due to MS".

Genetic factors, microbial and viral infections, smoking, serum vitamin D levels, obesity and nutritional habits are effective in the development of MS. Although the immune system seems to have a major effect on protection from MS, it is stated that the innate or acquired immune system may be effective in the development and occurrence of the disease. Although the mechanism is not clearly explained, it is stated that the disease may develop due to an autoimmune response that occurs as a result of damage to the blood-brain barrier caused by antigens formed against neurodegenerative diseases such as Alzheimer's or any viral infection.

MS is more common and economically burdensome in high-income countries such as Western Europe and North America, which are farthest from the equator. It is known that Western-style nutrition is dominant in these countries and that there is insufficient exposure to sunlight. The average age of onset of the disease has been determined as 32. Although it is more common in young adults and women, the female/male patient ratio has been reported to be between 1.5:1 and 2.5:1. It is estimated that there are 70 thousand MS patients in Turkey. It is known that approximately 2.8 million people have MS worldwide. The prevalence of the disease is determined as 35.9 MS patients per 100,000 people.

There is currently no known definitive treatment for the disease. However, disease-modifying treatments (DMTs) such as interferon beta-1a, interferon beta-1b, peginterferon beta-1a, glatiramer acetate, dimethyl fumarate, teriflunomide, natalizumab, fingolimod, cladribine, ocrelizumab and alemtuzumab are used to control the frequency of relapses, disability and progression of symptoms. Lifestyle changes applied in addition to DMTs can also improve the course of the disease. The aim of lifestyle changes applied to MS patients is to improve quality of life, reduce perceived fatigue and disability, and help improve the effects of brain fog that has come to the fore after the Covid-19 outbreak.

It has been determined that individuals diagnosed with MS change their nutritional behaviors, follow a diet rich in complex carbohydrates, low in simple sugar, saturated fat, gluten, and animal-based milk, and frequently use vitamin D supplements. Among the dietary models specifically applied for MS patients, the Best Bet diet, Overcoming MS (OMS), modified Paleolithic diet (Wahls diet), Swank diet, and McDougall diet are frequently emphasized in the literature. Apart from these, other dietary models applied to MS patients include anti-inflammatory diet, Mediterranean diet, Mediterranean- Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet, ketogenic diet, gluten-free diet, intermittent fasting and calorie-restricted diet models.

It is suggested that the MIND diet, developed by Rush University nutritional epidemiologist Martha Clare Morris and combining the Mediterranean diet with the DASH guidelines, may be effective in reducing the risk of developing neurodegenerative diseases (HARVARD MEDICAL SCHOOL Best Diets for Cognitive Fitness Foods). It has been shown that the MIND diet can improve cognitive functions and depression. Unlike the Mediterranean diet, the MIND diet is a dietary model that increases the consumption of fruits and green leafy vegetables and limits the consumption of cheese. The MIND diet consists of 15 components. 10 of the components (olive oil, oilseeds, green leafy vegetables, cooked vegetables, whole grains, legumes, fruit, poultry, seafood and red wine) are considered healthy for the brain, while 5 (red meat, butter, cheese, fast food, bakery products) are considered unhealthy. The European Society of Clinical Nutrition and Metabolism (ESPEN) recommends a diet rich in mono- and polyunsaturated fatty acids, limited to saturated fats, in its report on clinical nutrition in neurology for MS patients. The MIND diet meets this recommendation.

There are many studies investigating the effects of the Mediterranean diet, a component of the MIND diet, on disease-related symptoms in individuals with MS. However, studies examining the effects of the MIND diet in individuals with MS are quite limited. The study evaluated the link between MS and adherence to the MIND diet, which was developed specifically to prevent cognitive decline, and 77 MS patients and 148 healthy volunteers. Adherence to the MIND diet was associated with a reduced risk of MS. It was determined that the consumption of green leafy vegetables, other vegetables and beans, which are components of the MIND diet, was significantly lower in MS patients, while the consumption of cheese, poultry, pastries and desserts, and fried/fast foods was significantly higher, and it was shown that a higher MIND diet score was statistically significantly associated with a reduced probability of MS. In a cross-sectional study, the MIND diet compliance score was positively associated with thalamic volume. According to the results of the cross-sectional and longitudinal study, it was determined that the MIND diet positively affected the physical quality of life and fatigue in MS patients.

In a systematic review and meta-analysis study conducted by Fotros et al (2024), it was determined that fruit and vegetable consumption, which is also recommended in the MIND diet, has a potential protective effect against MS disease. It has been reported that a higher intake of plant protein, a component of the MIND diet, compared to animal protein, can reduce the symptoms and relapse rate of MS. According to the results of a retrospective study, fatty foods, snacks, sugary foods, fried and fast-food foods, which are among the components of the MIND diet and are in the group of unhealthy foods for the brain, are associated with the onset and development of MS, while reduced fruit consumption is associated with increased disability.

MS patients experience significant anxiety and problems regarding nutrition in the period after diagnosis. Many randomized controlled trials examining the dietary models and nutritional strategies applied by MS patients have emerged through literature review. When the relevant literature was examined, cross-sectional, prospective and retrospective studies investigating the effects of the MIND diet in MS patients were found, but no randomized controlled trial was found. This planned study is unique in that it is the first study to investigate the effects of the MIND diet on fatigue, quality of life and brain fog in MS patients using a parallel-design randomized controlled trial method. Based on this point, the study aims to evaluate the effects of the MIND diet on fatigue, quality of life, cognitive function, mental health and brain fog in MS patients.

With the results of this study; It will be possible to provide evidence on the subject to the international literature by determining the effect of the MIND diet applied to MS patients in Turkey on fatigue, quality of life, cognitive function, mental health and brain fog. Determining the positive effect of the MIND diet on the symptoms that develop due to possible MS disease and recommending this diet model to patients is important in terms of improving general health status and social life.

The hypotheses of the study; H0a: The quality of life health status parameter of the MIND diet applied to MS patients is similar to the control group.

H1a: The quality of life health status parameter of the MIND diet applied to MS patients is not similar to the control group.

H0b: The effect of the MIND diet applied to MS patients on fatigue is similar to the control group.

H1b: The effect of the MIND diet applied to MS patients on fatigue is not similar to the control group.

H0c: The effect of the MIND diet applied to MS patients on cognitive function is similar to the control group.

H1c: The effect of the MIND diet applied to MS patients on cognitive function is not similar to the control group.

H0d: The effect of the MIND diet applied to MS patients on mental health is similar to the control group.

H1d: The effect of the MIND diet applied to MS patients on mental health is not similar to the control group.

H0e: The effect of the MIND diet applied to MS patients on brain fog is similar to the control group.

H1e: The effect of the MIND diet on brain fog in MS patients is not similar to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult MS patients between the ages of 18-65 diagnosed according to the 2017 McDonald criteria
* Having been diagnosed with MS at least three months ago; patients are called for routine check-ups in the first and third months after starting treatment, as liver function tests and/or hemogram values may be impaired due to the treatment they started when they are newly diagnosed with MS. For this reason, it was planned to include patients whose check-ups were completed and no unexpected changes were observed in the blood parameters table due to the medication.
* No DMT change in the last 6 months
* Patients who use their medications regularly
* Not using nutritional support or supplements
* Patients with an EDSS score of ≤6
* Patients with a body mass index (BMI) between 18.5-24.9 kg/m2

Exclusion Criteria:

* MS patients who are pregnant or lactating
* Having another chronic metabolic disease and/or having had surgery in the last 3 months
* MS patients with limb deficiency
* MS patients on a special diet
* Patients using antidepressants and/or mood stabilizers
* Having had an attack and/or receiving steroid treatment in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-12-27 (Actual)

PRIMARY OUTCOMES:
The Effect of the MIND Diet on Quality of Life | 12 weeks from the start of the intervention
  -Multiple Sclerosis Quality of Life-54 Questionnaire consists of 12 subscales (I-Physical Health, II-Role limitations due to physical problems, III-Role limitations due to emotional problems, IV-Emotional well-being, V-Energy/fatigue, VI-Health perceptions, VII-Social functioning, VIII-Cognitive functioning, IX-Health distress, X-Sexual functioning, XI-Changes in health, XII-General quality of life). The scores of each subscale range from 0 to 100, with higher scores indicating better quality of life. MIND will be used to evaluate the role of the dietary intervention on quality of life.
Effect of the MIND diet on fatigue in MS patients | 12 weeks from the start of the intervention
  -Modified Fatigue Impact Scale, total score ranges from 0-84. Increasing score is associated with increased fatigue. It will be used to evaluate the role of MIND diet intervention on fatigue.
The effect of the MIND diet on brain fog in MS patients | 12 weeks from the start of the intervention
  -Brain Fog Scale, total score ranges from 30-150. An increase in score indicates an increase in brain fog level. It will be used to evaluate the effect of MIND diet on brain fog.

SECONDARY OUTCOMES:
The effect of the MIND diet on blood parameters | At the end of 12 weeks after the start of the intervention
  It will be determined whether the MIND diet has an effect on hemogram, biochemical parameters, folate, B12, D vitamins, C-reactive protein and thyroid hormones, including T3, T4 and TSH.
Effect of the applied MIND diet on body composition | After 12 weeks of MIND diet or healthy eating program application
  The neck, waist and hip circumference measurements will be made in cm. The data collected will determine the change in the body composition of the individuals and which body tissue this change is due to (thanks to the circumference measurements it is due to the change in fat or muscle mass).

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University/Muğla Training and Research Hospital Neurology Polyclinic, Muğla, Mentese, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The planned study is original in that it is the first study to investigate the effect of the MIND diet applied to MS patients on fatigue, quality of life and brain fog using a parallel-design randomized controlled trial method. Based on this point, this thesis aims to evaluate the effect of the MIND diet applied to MS patients on fatigue, quality of life, cognitive function, mental health and brain fog. With the results of this study; It will be possible to provide evidence on the subject to the international literature by determining the effect of the MIND diet applied to MS patients in Turkey on fatigue, quality of life, cognitive function, mental health and brain fog. Determining the positive effect of the MIND diet on symptoms developing due to possible MS disease and recommending this diet model to patients is important in terms of improving general health status and social life.
Supporting Information: Study Protocol, SAP, CSR